CLINICAL TRIAL: NCT03278509
Title: Randomized Evaluation of Decreased Usage of betablocCkErs After Myocardial Infarction in the SWEDEHEART Registry - A Registry-based, Randomized, Parallel, Open-label, Multicenter Trial (REDUCE-SWEDEHEART)
Brief Title: Evaluation of Decreased Usage of Betablockers After Myocardial Infarction in the SWEDEHEART Registry (REDUCE-SWEDEHEART)
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Uppsala University (Other); The Swedish Research Council (Other Government)
Responsible Party: Principal Investigator, Dr. Tomas Jernberg, Co-ordinating principal investigator, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EudraCT number 2017-002336-17
Record Dates: First submitted 2017-08-31; First posted 2017-09-11 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Acute Myocardial Infarction; Non-ST Elevation Myocardial Infarction; ST Elevation Myocardial Infarction
MeSH Terms: conditions — Non-ST Elevated Myocardial Infarction; ST Elevation Myocardial Infarction | interventions — Metoprolol; Bisoprolol

STUDY DESIGN:
Intervention Model Description: A registry-based, randomized, parallel, open-label, multicenter trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Oral beta-blocker treatment (Experimental): Patients randomized to beta-blockade will be prescribed oral beta-blocker (metoprolol succinate or bisoprolol) at a dose according to the treating physician. Metoprolol succinate will be strongly recommended as first choice. Bisoprolol will be allowed as an alternative. Atenolol (or any other beta-blocker therapy) will not be allowed. The treating physician will be encouraged to aim for a dose of ≥ 100 mg for metoprolol succinate and ≥ 5 mg for bisoprolol. Prescribed treatment and dosing will be registered. Initiation (whether the prescribed drug is dispensed) and adherence (defined as proportion of prescribed tablets that are dispensed), and persistence (time on treatment) will also be recorded via the Drug prescription registry.
  Interventions: Drug: Metoprolol Succinate; Drug: Bisoprolol
- No beta-blocker treatment (No Intervention): Patients randomized to no beta-blockade will be discouraged to use beta-blockade as long as there is no other indication than strictly secondary prevention after myocardial infarction. Patients assigned to no beta-blockade also receive best evidence-based care, without beta-blockers. For blood pressure control, other drugs than beta-blockers will be recommended as first-line treatment. Regarding later use of beta-blockade, follow up is performed in the Drug prescription registry. Patients will be asked to provide future physicians with the written information about the study when beta-blockade treatment is discussed.

INTERVENTIONS:
Drug: Metoprolol Succinate — Eligible patients randomized to active treatment will receive long-term oral beta-blockade (metoprolol succinate or bisoprolol).
  Arms: Oral beta-blocker treatment
Drug: Bisoprolol — Please see the section above.
  Arms: Oral beta-blocker treatment

SUMMARY:
Long-term beta-blocker therapy has not been investigated in contemporary randomized clinical trials in patients with myocardial infarction and normal heart function. The aim of this study is to determine whether long-term treatment with oral beta-blockade in patients with myocardial infarction and preserved left ventricular systolic ejection fraction reduces the composite of death of any cause or new myocardial infarction..

DETAILED DESCRIPTION:
REDUCE-SWEDEHEART is designed as a registry-based, randomized, parallel, open-label, multicenter trial.

Patients, day 1-7 after myocardial infarction, who have undergone a coronary angiography and with preserved left ventricular systolic ejection fraction will be randomized to either oral beta-blockade (see "Intervention" for detailed description) at a dose according to the treating physician, or no beta-blockade. To allow quick inclusion the randomization module will be accessible by a simple web-based log-in procedure. Concomitantly, all baseline data about each individual patient will be collected from the SWEDEHEART registry. Patients will then be followed regarding all-cause mortality, myocardial infarction, heart failure, atrial fibrillation, and patient-related outcome measures (for a subgroup of patients). Patients that are eligible but not included in REDUCE-SWEDEHEART will also be followed regarding chosen treatment and the primary and secondary endpoints.

Follow-up will continue until 379 primary endpoints have been observed (endpoint driven). All analyses will be performed on the intention-to-treat set, defined as all intentionally randomized patients, by randomized treatment. The primary endpoint is death or new MI. Information about death will be obtained from the Swedish population registry. Information regarding new myocardial infarction during hospitalization and readmission because of myocardial infarction or other outcome (secondary outcomes, see section below), will be obtained from the SWEDEHEART-registry (for myocardial infarction) and the patient registry of the National board of health and welfare.

ELIGIBILITY:
Inclusion Criteria:

1. Age≥18 years.
2. Day 1-7 after MI as defined by the universal definition of MI, type 1, included in the SWEDEHEART registry.
3. Undergone coronary angiography during hospitalization.
4. Obstructive coronary artery disease documented by coronary angiography, i.e. stenosis ≥ 50 %, FFR ≤ 0.80 or iFR ≤ 0.89 in any segment at any time point before randomization.
5. Echocardiography performed after the MI showing a normal ejection fraction (EF≥50%).
6. Written informed consent obtained.

Exclusion Criteria:

1. Any condition that may influence the patient's ability to comply with study protocol.
2. Contraindications for beta-blockade
3. Indication for beta-blockade other than as secondary prevention according to the treating physician.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5000 (Estimated)
Dates: Start 2017-09-11 (Actual); Primary Completion 2023-11-16 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Time to the composite of death of any cause or MI | through study completion, an average of 3 year
  Time to the composite of death of any cause or MI on an intention to treat basis (ITT)

SECONDARY OUTCOMES:
All-cause death | through study completion, an average of 3 year
  Time to the individual component of the primary endpoint of any cause of death.
Myocardial infarction | through study completion, an average of 3 year
  Time to the individual component of the primary endpoint of MI.
Cardiovascular death | through study completion, an average of 3 year
  Time to cardiovascular death.
Heart failure | through study completion, an average of 3 year
  Time to hospital readmission due to heart failure (primary [main] diagnosis)
Atrial fibrillation | through study completion, an average of 3 year
  Time to hospital readmission due to atrial fibrillation (primary [main] diagnosis)
Bradycardia, Advanced AV-block, hypotension, syncope or need for pacemaker | through study completion, an average of 3 year
  Time to hospital readmission due to bradycardia or advanced AV-block or hypotension or syncope or need for pacemaker (primary [main] diagnosis)
Asthma or Chronic Obstructive Pulmonary Disease | through study completion, an average of 3 year
  Time to hospital readmission due to asthma or chronic obstructive pulmonary disease (primary [main] diagnosis)
Stroke | through study completion, an average of 3 year
  Time to hospital readmission due to stroke (primary [main] diagnosis)
Health related quality of life (HRQOL) | Estimated maximal follow-up for each patient for this outcome is 1 year.
  Health related quality of life (HRQOL) measured by EQ-5D in patients younger than 75 years of age
Health care costs | through study completion, an average of 3 year
  Health care cost analysis concerning the use beta-blocker treatment

OTHER OUTCOMES:
Anxiety and depression | 8 weeks and 12 months after randomization
  Anxiety and depression measured by Hospital Anxiety and Depression Scale (HADS)
Wellbeing | 8 weeks and 12 months after randomization
  Wellbeing measured by WHO-5 Wellbeing Index
Cardiac Anxiety | 8 weeks and 12 months after randomization
  Cardiac Anxiety measured by Cardiac Anxiety Questionnaire (CAQ)
Sexual function | 8 weeks and 12 months after randomization
  Sexual function measured by Arizona Sexual Experiences Scale (ASEX)

CONTACTS AND LOCATIONS:
Overall Officials: Tomas Jernberg, MD PhD, Principal Investigator — Karolinska Institutet; Bertil Lindahl, MD PhD, Study Chair — Uppsala, Clinical Sciences
Locations (1):
- Danderyd Hospital, Cardiac Intensive Care, Danderyd, Stockholm County, Sweden

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Leissner P, Johansson M, Mars K, Held C, Hofmann R, Olsson EMG. Psychometric properties of the Swedish cardiac anxiety questionnaire: a Rasch analysis. Sci Rep. 2025 Nov 24;15(1):41834. doi: 10.1038/s41598-025-28073-8. PMID 41286053
- [Derived] Leening MJG, Boersma E. The perpetual need of randomized clinical trials: challenges and uncertainties in emulating the REDUCE-AMI trial. Eur J Epidemiol. 2024 Apr;39(4):343-347. doi: 10.1007/s10654-024-01127-3. Epub 2024 May 11. PMID 38733447
- [Derived] Matthews AA, Dahebreh IJ, MacDonald CJ, Lindahl B, Hofmann R, Erlinge D, Yndigegn T, Berglund A, Jernberg T, Hernan MA. Prospective benchmarking of an observational analysis in the SWEDEHEART registry against the REDUCE-AMI randomized trial. Eur J Epidemiol. 2024 Apr;39(4):349-361. doi: 10.1007/s10654-024-01119-3. Epub 2024 May 8. PMID 38717556
- [Derived] Yndigegn T, Lindahl B, Mars K, Alfredsson J, Benatar J, Brandin L, Erlinge D, Hallen O, Held C, Hjalmarsson P, Johansson P, Karlstrom P, Kellerth T, Marandi T, Ravn-Fischer A, Sundstrom J, Ostlund O, Hofmann R, Jernberg T; REDUCE-AMI Investigators. Beta-Blockers after Myocardial Infarction and Preserved Ejection Fraction. N Engl J Med. 2024 Apr 18;390(15):1372-1381. doi: 10.1056/NEJMoa2401479. Epub 2024 Apr 7. PMID 38587241
- [Derived] Humphries S, Mars K, Hofmann R, Held C, Olsson EMG. Randomized evaluation of routine beta-blocker therapy after myocardial infarction quality of life (RQoL): design and rationale of a multicentre, prospective, randomized, open, blinded endpoint study. Eur Heart J Open. 2023 Apr 10;3(3):oead036. doi: 10.1093/ehjopen/oead036. eCollection 2023 May. PMID 37265820
- [Derived] Granger CB, Pocock SJ, Gersh BJ. The need for new clinical trials of old cardiovascular drugs. Nat Rev Cardiol. 2023 Feb;20(2):71-72. doi: 10.1038/s41569-022-00819-1. No abstract available. PMID 36526898